CLINICAL TRIAL: NCT02727426
Title: Influence of High Salt Diet on Microvascular Reactivity in Young Healthy Subjects
Brief Title: Dietary Salt and Microvascular Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Principal Investigator, Ines Drenjancevic, Vice Dean for Science, Faculty of Medicine Josip Juraj Strossmayer University of Osijek, Josip Juraj Strossmayer University of Osijek
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 215861071012
Record Dates: First submitted 2016-03-15; First posted 2016-04-04 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: Salt; Excess
Keywords: microvascular function; laser Doppler flowmetry; high salt diet
MeSH Terms: interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- low salt diet (Experimental): All subjects will be instructed to maintain a low-sodium (LS) diet, with an intake of less than 2.3 g of salt per day (DASH eating plan; US Department of Health and Human Services, 2006) for 7 days (washout period).
  Interventions: Other: Low Salt (LS) diet
- high salt diet (Experimental): After washout period, all subjects will be instructed to maintain a high-sodium (HS) diet, with an intake of 11.2 g of salt per day for 7 days.
  Interventions: Other: High Salt (HS) diet

INTERVENTIONS:
Other: Low Salt (LS) diet — Intake of less than 2.3 g of salt per day for 7 days.
  Arms: low salt diet
Other: High Salt (HS) diet — Intake of 11.2 g of salt per day for 7 days.
  Arms: high salt diet

SUMMARY:
It is well accepted that high-salt (HS) intake is an essential risk factor in development and progression of hypertension. Results of some recent studies suggest that some of the deleterious effects of a HS diet are independent of elevated blood pressure (BP) and may occur in normotensive individuals and are associated with impaired endothelial function. However, the effects of acute salt loading on endothelial function and vascular reactivity in young healthy individuals are still scarce and inconsistent.

The purpose of present study is to determine whether one week of HS intake affects microvascular reactivity in young healthy subjects without changes in BP. In addition, the investigators sought to evaluate if potential HS diet-induced microvascular dysfunction is associated with changes in oxidative stress level and/or with modification of immunological response in young healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

- healthy volunteers

Exclusion Criteria:

* oral contraceptives
* drugs that could affect the endothelium
* hypertension
* coronary artery disease
* diabetes
* hyperlipidaemia
* renal impairment
* cerebrovascular and peripheral artery disease

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-05 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
microvascular reactivity | two weeks after starting the protocol
  Cutaneous microvascular blood flow will be measured by Laser Doppler Flowmetry in response to vascular occlusion (post occlusive reactive hyperemia- PORH) and in response to iontophoresis of acetylcholine (ACh) (endothelium dependent vasodilation) before and after diet protocols.

SECONDARY OUTCOMES:
oxidative stress | two weeks after starting the protocol
  As direct indicator of oxidative stress, byproducts of lipid peroxidation - TBARS method (Thiobarbituric Acid Reactive Substances) with malondialdehyde (MDA) as standard (µM MDA) will be measured before and after LS and HS diet protocol (spectrophotometric method).
modification of immunological response by high salt diet | two weeks after starting the protocol
  Activated monocytes/macrophages and neutrophils will be measured by flow cytometry, with distinction of subpopulation of monocytes/macrophages (classical/nonclassical), their activation and the expression of the integrin LFA-1 (lymphocyte function-associated antigen 1) and VLA-4 (Very Late Antigen-4) - ligands VCAM-1 (vascular cell adhesion molecule 1 ) and ICAM-1 (vascular cell adhesion molecule 1).
antioxidant capacity | two weeks after starting the protocol
  As an indicator of antioxidant capacity, the ferric reducing ability of plasma - the FRAP assay (Ferric reducing ability of plasma) with Trolox used as standard (mM Trolox) will be measured before and after LS and HS diet protocol (spectrophotometric method).

CONTACTS AND LOCATIONS:
Overall Officials: Ines Drenjancevic, MD, PhD, Principal Investigator — Faculty of Medicine, University of Osijek, Croatia
Locations (1):
- Faculty of Medicine Osijek, Laboratory for Clinical and Sport Physiology, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cavka A, Cosic A, Jukic I, Jelakovic B, Lombard JH, Phillips SA, Seric V, Mihaljevic I, Drenjancevic I. The role of cyclo-oxygenase-1 in high-salt diet-induced microvascular dysfunction in humans. J Physiol. 2015 Dec 15;593(24):5313-24. doi: 10.1113/JP271631. Epub 2015 Dec 7. PMID 26498129
- [Background] Cavka A, Cosic A, Grizelj I, Koller A, Jelakovic B, Lombard JH, Phillips SA, Drenjancevic I. Effects of AT1 receptor blockade on plasma thromboxane A2 (TXA2) level and skin microcirculation in young healthy women on low salt diet. Kidney Blood Press Res. 2013;37(4-5):432-42. doi: 10.1159/000355723. Epub 2013 Oct 13. PMID 24247418
- [Background] Cavka A, Jukic I, Ali M, Goslawski M, Bian JT, Wang E, Drenjancevic I, Phillips SA. Short-term high salt intake reduces brachial artery and microvascular function in the absence of changes in blood pressure. J Hypertens. 2016 Apr;34(4):676-84. doi: 10.1097/HJH.0000000000000852. PMID 26848993